CLINICAL TRIAL: NCT06856382
Title: Identification of Paraneoplastic and Intratumor Microplastics in Gastric Cancer and Their Association Analysis With Macrogenomics and Metabolomics
Brief Title: The Association Between Microplastics and Macrogenomics and Metabolomics in Gastric Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Dong Peng (Other)
Responsible Party: Sponsor-Investigator, Dong Peng, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 2024-530-01
Record Dates: First submitted 2025-02-25; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cancers
Keywords: Gastric cancer; Microplastics; Macrogenomic; Metabolomics; Microenvironment
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — surgically resected tissue and serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- the gastric cancer group: patients diagnosed with gastric cancer
  Interventions: Diagnostic Test: gastric cancer

INTERVENTIONS:
Diagnostic Test: gastric cancer — Patients diagnosed with gastric cancer by pathological biopsy.

SUMMARY:
The aim of this study was to identify and quantify microplastics in blood, stool, and tumor surgical specimens from gastric cancer patients by analyzing the nature, type, and abundance of microplastics using laser direct infrared (LDIR) spectroscopy, scanning electron microscopy (SEM), and pyrolysis-gas chromatography-mass spectrometry (Py-GC/MS). Meanwhile, combining macro-genomic and metabolomic techniques to explore the association between microplastics and host microbiota and metabolic profiles, and to reveal the potential effects of microplastics on gastric cancer incidence and development will provide new insights into the relationship between microplastic contamination and gastric cancer, as well as an important scientific basis for future public health strategies and cancer prevention and control measures.

DETAILED DESCRIPTION:
This This study is planned to collect blood, cancer and paracancer tissues, and stool samples from 20 patients with gastric cancer, 2 gastric cancer tissues (at least 1cm^3 each), 2 gastric paracancer tissues (at least 1cm^3 each), 2 venous bloods (5ml each), and 1 stool (at least 10g each) from each patient. Samples will be collected from December 2024 through November 2025, with an expected total of 140 samples. Sample collection, transportation, and storage are described in IV.2. & 3. Samples will be analyzed for the type, nature, and abundance of microplastics by Laser Direct Infrared Spectroscopy (LDIR), Scanning Electron Microscopy (SEM), and Pyrolysis-Gas Chromatography-Mass Spectrometry (Py-GC/MS), which is expected to detect microplastics such as polyamides, polyethylene terephthalate (PET), and polyvinyl chloride (PVC). At the same time, blood and tissue samples will be metabolomically assayed using NNR-IVD technology and macro-genomic sequencing will be performed to explore potential associations between microplastics and microbiota and metabolic pathways in gastric cancer patients. By analyzing the distribution characteristics of microplastics in gastric cancer patients and their relationship with microbial communities and metabolic pathways, this study will reveal the impact of microplastics on the tumor microenvironment and further understand their role in gastric cancer development and progression.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years old;
* diagnosed with gastric cancer by pathology before surgery and not receiving chemotherapy, radiotherapy or immunotherapy;
* no history of other gastrointestinal diseases;
* complete clinical data and basic information;
* willing to participate in this study and sign an informed consent form.

Exclusion Criteria:

* Patients receiving neoadjuvant radiotherapy or chemotherapy;
* patients with other malignant tumors other than gastric cancer;
* patients with incomplete or unclear pathological data;
* individuals who are not willing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with colorectal cancer by pathological biopsy were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Types of microplastics in gastric cancerous and paracancerous tissues (categorical measure) | The date of microplastics testing, assessed up to 1 week after surgery.
  Polymer types of microplastics in gastric tissues Time Frame: Intraoperative sampling Measuring tool: μ-FTIR spectroscopy Unit: Categorical classification (e.g., polyethylene, polypropylene, etc.)

SECONDARY OUTCOMES:
Physical-chemical properties of microplastics in gastric cancerous and paracancerous tissues (continuous measure) | The date of microplastics testing, assessed up to 1 week after surgery.
  Morphological characteristics of microplastics in gastric tissues Time Frame: Intraoperative sampling Measuring tool: Optical microscopy Unit: Size (μm), shape distribution (%)
Abundance of microplastics in gastric cancerous and paracancerous tissues (count/particles per gram) | The date of microplastics testing, assessed up to 1 week after surgery.
  Microplastic abundance in gastric tissues Time Frame: Intraoperative sampling Measuring tool: Gravimetric analysis/particle counting Unit: Particles per gram tissue

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data sharing is not permitted by the Ethics Committee of the First Affiliated Hospital of Chongqing Medical University.